CLINICAL TRIAL: NCT00251381
Title: Open Label Randomized Phase II, Multicentre, Pilot Study to Evaluate Safety and Efficacy of the Combination of Cetuximab and Concomitant-Boost Accelerated Radiotherapy Followed or Not by a Complementary Treatment With Cetuximab in Patients With Locally Advanced Oropharynx Squamous Cell Carcinoma.
Brief Title: Cetuximab & Concomitant-Boost Accelerated RT in Patients With Locally Advanced Oropharynx Squamous Cell Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trial Form Support S.L. (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62202-655
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Oropharyngeal Neoplasms
Keywords: Oropharyngeal Neoplasms; Cetuximab; Concomitant-boost accelerated radiotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Cetuximab

INTERVENTIONS:
Drug: Cetuximab

SUMMARY:
The purpose of this study is to determine the 1-year rate of locoregional disease control in the experimental arm, using a control arm to avoid selection bias.

DETAILED DESCRIPTION:
* To determine the 1-year rate of locoregional disease control in the experimental arm, using a control arm to avoid selection bias.
* To determine the 2 and 3 year rate of locoregional disease control.
* To evaluate the safety and toxicity of the combination of cetuximab and concomitant-boost accelerated radiotherapy followed by 12 weeks of complementary treatment with cetuximab. Both acute and chronic toxicity will be assessed.
* To determine specific disease-free survival, event-free survival, disease-specific survival and overall survival
* To determine acute and late toxicity
* To determine EGFR, p53, Ki67, and evaluate its value as a prognostic factor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Aged between 18 and 80, inclusive.
* Karnofsky functional status >= 70% at the time of enrolment in study.
* Life expectancy of more than 3 months.
* Histologically confirmed diagnosis of oropharyngeal squamous cell carcinoma: base of tongue, vallecula, tonsil and tonsillar fossa and pillars, glossotonsillar sulcus, inferior surface of the soft palate, uvula and lateral and posterior oropharyngeal wall.
* Stage III or IV with no evidence of distant metastasis (IVA or IV B)
* Patients in medical conditions to receive a radical concomitant-boost accelerated radiotherapy treatment.
* Neutrophils >= 1500/ mm3, platelet count >= 100 000/ mm3 and haemoglobin >= 10 g/ dL.
* Proper liver function: total bilirubin <= 1.5 x upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 x ULN.
* Proper renal function: serum creatinine <= 1.5 x ULN; if the values are > 1.5 x ULN, creatinine clearance should be >= 55 ml/min.
* Serum calcium within normal limits.
* Adequate nutritional state: weight loss < 20% with respect to usual weight and serum albumin > 35 g/l.
* Effective birth control method if there is possibility of conception and/or pregnancy.
* Availability of tumour tissue for immunohistochemical analysis of EGFR expression.

Exclusion Criteria:

* Metastatic disease.
* Previous surgical, radiotherapy and/or chemotherapy treatment for the disease in the study.
* Other non-oropharyngeal tumour sites in the head and neck area.
* Other previous and/or simultaneous squamous cell carcinoma.
* Diagnosis of any other cancer in the previous 5 years, except properly treated carcinoma in situ of the uterine cervix and/or basal cell skin carcinoma.
* Active infection (infection requiring intravenous antibiotics), including active tuberculosis and diagnosed HIV.
* Uncontrolled hypertension defined as systolic blood pressure >= 180 mm Hg and/or diastolic blood pressure >= 130 mm Hg at rest.
* Pregnancy (absence of pregnancy must be confirmed with the serum-HCG test) or breast-feeding women.
* Chronic, concomitant systemic immunotherapy, or hormonal treatment for the cancer.
* Other concomitant anti-cancer treatments.
* Clinically significant coronary artery disease, history of myocardial infarction in the previous 12 months or high risk of out of control arrhythmia or cardiac insufficiency.
* Chronic obstructive pulmonary disease which may have required > 3 hospitalisations in the previous 12 months.
* Out of control active peptic ulcer.
* Presence of a psychological or medical illness which might impede the patient from carrying out the study or giving his or her signature on the informed consent
* Known drug abuse (with the exception of excessive alcohol consumption)
* Known allergic reaction to any of the components of the treatment to be studied.
* Previous treatment with monoclonal antibodies or signal transduction inhibitors or other EGFR-targeted treatment.
* Any experimental treatment in the 30 days prior to enrolment in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-11; Study Completion 2009-11

PRIMARY OUTCOMES:
1-year rate of Locoregional Disease Control in the experimental arm, deffined as complete and persistent disappearance of disease in the primary tumour and regional lymph nodes.

SECONDARY OUTCOMES:
Toxicity and safety of treatment will be evaluated using the Common Toxicity Criteria (CTC) of the NCI, version 3.0.; and late toxicity from radiotherapy, using RTOG/EORTC Late Radiation Morbidity Scoring Scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Mesia, MD, Principal Investigator — Institut Catala Oncologia: Hospital Durán y Reynals; Joaquin Gomez, MD, Principal Investigator — Institut Catala Oncologia: Hospital Durán y Reynals
Locations (18):
- Spain (18):
  - Hospital Germans Tries i Pujol, Badalona, Barcelona
  - H. del Mar / H. de la Esperanza, Barcelona, Barcelona
  - H. de la Santa Creu I Sant Pau, Barcelona, Barcelona
  - Institut Catala Oncologia: Hospital Duran y Reynals, L'Hospitalet de Llobregat, Barcelona
  - Centro Oncológico Regional de Galicia, A Coruña, Coruña
  - H. Josep Trueta (ICO), Girona, Girona
  - H. G. Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Clinica Ruber Internacional, Madrid, Madrid
  - H. Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - H. Gregorio Marañón, Madrid, Madrid
  - Complejo Hospitalario Virgen de la Victoria, Málaga, Malaga
  - H. Carlos Haya, Málaga, Malaga
  - H.U. Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - H. U. de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - H. do Meixoeiro, Vigo, Vigo
  - H.U. de Santiago, Santiago